CLINICAL TRIAL: NCT05512494
Title: A Randomized, Double-blind Clinical Trial to Evaluate Lot-to-lot Consistency , Immunogenicity and Safety of Quadrivalent Influenza Vaccine (Split Virion), Inactivated in Health Populations Aged 9~59 Years Old
Brief Title: Lot-to-lot Consistency of Quadrivalent Influenza Vaccine (Split Virion), Inactivated
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO-QINF-4003
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-07

CONDITIONS: Seasonal Influenza
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadrivalent Influenza Vaccine (Split Virion), inactivated Lot 1 (Experimental): 420 participants including 120 subjects aged 9-17 years and 300 subjects aged 18-59 years will receive one dose of quadrivalent influenza vaccine of commercial scale production lot 1.
  Interventions: Biological: Quadrivalent Influenza Vaccine (Split Virion), inactivated
- Quadrivalent Influenza Vaccine (Split Virion), inactivated Lot 2 (Experimental): 420 participants including 120 subjects aged 9-17 years and 300 subjects aged 18-59 years will receive one dose of quadrivalent influenza vaccine of commercial scale production lot 2.
  Interventions: Biological: Quadrivalent Influenza Vaccine (Split Virion), inactivated
- Quadrivalent Influenza Vaccine (Split Virion), inactivated Lot 3 (Experimental): 420 participants including 120 subjects aged 9-17 years and 300 subjects aged 18-59 years will receive one dose of quadrivalent influenza vaccine of commercial scale production lot 3.
  Interventions: Biological: Quadrivalent Influenza Vaccine (Split Virion), inactivated

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine (Split Virion), inactivated — The Quadrivalent Influenza Vaccine manufactured by Sinovac Biotech Co.,Ltd. The four influenza strains（including 4 antigens H1N1, H3N2, BV and BY, 15μg for each) in 0.5 mL of sodium chloride,disodium hydrogen phosphate,sodium dihydrogen phosphate water for per injection.The routine of administration is intramuscular injection into deltoid region.And the immunization schedule is one dose of quadrivalent influenza vaccine on day 0.

SUMMARY:
This study is a randomized, double-blind phase Ⅳ clinical trial of quadrivalent influenza vaccine (Split Virion), inactivated manufactured by Sinovac Biotech Co., Ltd.The purpose of this study is to evaluate the lot-to-lot consistency, immunogenicity and safety of quadrivalent influenza vaccine (Split Virion), inactivated in health subjects aged 9-59 years old.

DETAILED DESCRIPTION:
This study is a randomized, double-blind phase Ⅳ clinical trial in health subjects aged 9-59 years old to evaluate the lot-to-lot consistency,immunogenicity and safety of quadrivalent influenza vaccine (Split Virion), inactivated.The experimental vaccine was manufactured by Sinovac Biotech Co., Ltd.A total of 1260 subjects,including 360 subjects aged 9-17 years and 900 subjects aged 18-59 years will be enrolled.The subjects in each age group will be randomly divided into three groups in a ratio of 1:1:1 to receive one dose of three lots of quadrivalent influenza vaccine (Split Virion), inactivated produced on a commercial scale,respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 9-59 years;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 9-17 years, both subjects and guardians need to sign the informed consent form).
* Proven legal identity.

Exclusion Criteria:

* Received seasonal influenza vaccine for 2022-2023 influenza season, or had an influenza vaccine schedule during the study;
* Suffering from seasonal influenza in the past 6 moths;
* Women of childbearing age (menarche to premenopause) are pregnant(including positive urine pregnancy test), breastfeeding or planning pregnancy within 1 month;
* Patients with fever on the day of vaccination,underarm body temperature>37.2 ℃;
* History of asthma, allergy to vaccines or vaccine components, and serious adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Severe chronic diseases,such as severe cardiovascular diseases, hypertension(Systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg) and diabetes that cannot be controlled by drugs, liver or kidney diseases,malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Autoimmune disease or immune deficiency/immunosuppression;
* Thyroid disease or history of thyroidectomy,absence of spleen, functional functional asplenia,and absence of spleen or splenectomy as a result of any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* A long history of alcohol or drug abuse;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs within 30 days prior to receiving the investigational vaccine;
* Receipt of attenuated live vaccines or COVID-19 vaccines in the past 14 days,receipt of inactivated or subunit vaccines in the past 7 days;
* The subjects participated in other clinical trials during the follow-up period or will be planned to participate other clinical trials during the follow-up period;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 9 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1260 (Actual)
Dates: Start 2022-11-27 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index of GMT | 28 days after vaccination
  GMT of HI antibodies of each influenza strain at 28 days after vaccination.

SECONDARY OUTCOMES:
Immunogenicity index of seroconversion rate | 28 days after vaccination
  Seroconversion rate of HI antibodies of each influenza strain at 28 days after vaccination.
Immunogenicity index of protection rate | 28 days after vaccination
  Protection rate of HI antibodies of each influenza strain at 28 days after vaccination (HI antibody titer ≥1:40).
Immunogenicity index of GMI | 28 days after vaccination
  GMI of HI antibodies of each influenza strain at 28 days after vaccination.
Safety index of the incidence of adverse reactions | From 0 to 28 days after vaccination.
  Incidence of adverse reactions from 0 to 28 days after vaccination.
Safety index -The incidence of adverse reactions | From 0 to 7 days after vaccination.
  Incidence of adverse reactions from 0 to 7 days after vaccination.
Safety index of the incidence of serious adverse events | From 0 to 28 days after vaccination
  Incidence of serious adverse events from 0 to 28 days after vaccination.
Safety index of incidence of adverse events | From 0 to 28 days after vaccination
  Incidence of adverse events of special concern from 0 to 28 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghu Guan, Principal Investigator — Guizhou Provincial Center for Disease Prevention and Control
Locations (1):
- Yuping Dong Autonomous County Center for Disease Control and Prevention, Zhumadian, Guizhou, China

REFERENCES:
- [Derived] Gao Y, Yang X, Li X, Chen H, Li Y, Tan X, Yu D, Feng T, Zhou S, Lei S, Zhao C, Wang J, Guan Q. Lot-to-lot consistency, immunogenicity and safety of a quadrivalent split virion inactivated influenza vaccine in healthy population aged 9-59 years: A randomized, double-blind, controlled, phase IV clinical trial. Vaccine. 2024 Aug 30;42(21):126182. doi: 10.1016/j.vaccine.2024.126182. Epub 2024 Aug 6. PMID 39116486